CLINICAL TRIAL: NCT05671640
Title: Feasibility Study of the DragonFly-T Transcatheter Tricuspid Valve Repair System for the Treatment of Tricuspid Regurgitation
Brief Title: Feasibility Study of the DragonFly-T System for Severe Tricuspid Regurgitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangzhou Valgen Medtech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DragonFly-T-2
Record Dates: First submitted 2022-12-20; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Tricuspid Regurgitation
Keywords: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DragonFly-T Transcatheter Tricuspid Valve Repair System (Experimental): The experimental group is allocated to use a novel tricuspid valve repair system for edge-to-edge repair manufactured by Hangzhou Valgen Medtech Co., Ltd.
  Interventions: Device: DragonFly-T Transcatheter Tricuspid Valve Repair System

INTERVENTIONS:
Device: DragonFly-T Transcatheter Tricuspid Valve Repair System — To conduct edge-to-edge repair with DragonFly-T System under the guidance of transesophageal echocardiography.

SUMMARY:
This study is a prospective design. Patients are severe tricuspid regurgitation (TR) (≥ 3+) who remained clinically symptomatic after guideline-directed medical treatment. After signing an informed consent form, subjects are enrolled and treated with the DragonFly-T Transcatheter Tricuspid Valve Repair System. All subjects receive clinical follow-up immediately after the procedure, before discharge, 30 days after the procedure, 6 months after the procedure, 12 months, and 2, 3, 4, and 5 years after the procedure.

The incidence of MAEs (Major Adverse Events) at 30 days is used as the safety endpoint. The MAEs include stroke, cardiovascular death, new renal failure, endocarditis requiring surgery, and non-elective cardiovascular interventions due to device-related adverse events.

The efficacy endpoints include acute procedural success, acute device success, the incidence of all-cause mortality and/or heart failure rehospitalization at 12 months after the procedure, the percentage of patients with tricuspid regurgitation of 2+ or less, the percentage of patients with tricuspid regurgitation reduced by at least one grade, the improvement in 6 minutes walk test, New York Heart Association (NYHA) class, quality of life change as assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ) score and change in edema scale grading.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. In the judgment of the local cardiac team, the patient has been adequately treated according to applicable standards (including medical management), including:

   1. Optimal pharmacological therapy for TR (e.g. diuretics);
   2. Drug and/or interventional treatment of mitral regurgitation, atrial fibrillation, coronary artery disease, and heart failure;
   3. The Eligibility Committee confirms that the patient has received adequate medical treatment.
3. Despite the drug optimization treatment according to the above method, patients still have symptoms of TR (TR grade≥3+).
4. New York Heart Association (NYHA) Cardiac function Class II-IVa.
5. The patient is suitable for transcatheter tricuspid valve repair, suitable for the use of the study device, and the femoral vein access is feasible and can accommodate a 24F catheter.
6. Patient must provide written informed consent before any steps related to the study.

Exclusion Criteria:

1. Tricuspid valve leaflet anatomy, which may preclude clip implantation or proper clip positioning on the leaflets, including but not limited to the following:

   1. Evidence of calcification in the grasping area;
   2. Presence of a severe coaptation defect of the tricuspid leaflets;
   3. Severe leaflet defect(s) and cleft preventing proper device placement determined by ECL;
   4. Epstein anomaly.
2. Previous tricuspid valve surgery or transcatheter therapy.
3. Echocardiography suggested intracardiac thrombus, tumor, or mass.
4. Transthoracic Echocardiogram and Transesophageal Echocardiography are unable to evaluate tricuspid valve anatomy.
5. Refractory heart failure requiring intervention (e.g., left ventricular assist device, heart transplantation) (ACC/AHA Stage D heart failure).
6. Severe and uncontrolled hypertension: systolic blood pressure ≥ 180mmHg and/or diastolic blood pressure ≥ 110mmHg.
7. Active endocarditis, active rheumatic heart disease, or rheumatic heart valvular disease leading to tricuspid valve leaf lesions (poor valve leaf compliance, perforation, etc.).
8. Had myocardial infarction or unstable angina within 4 weeks; Untreated severe coronary artery stenosis requiring revascularization.
9. Percutaneous coronary intervention was performed within 30 days before surgery, except for coronary angiography.
10. Hemodynamic instability, defined as systolic blood pressure < 90mmHg, with or without cardiogenic shock, or requiring intra-aortic balloon counterpulsation or other hemodynamic support devices.
11. Bleeding diseases or coagulation disorders, or antithrombotic drug therapy contraindications.
12. Acute peptic ulcer or gastrointestinal bleeding within 3 months before surgery.
13. Severe cirrhosis (Child's grade C).
14. Allergy to the device material.
15. Life expectancy of fewer than 12 months.
16. Women who are pregnant, breastfeeding, or planning to become pregnant.
17. Participated in any drug and/or medical device clinical trials within 1 month prior to the trial.
18. The researchers do not consider it appropriate to be enrolled in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-02-10 (Estimated); Study Completion 2024-01-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse events (MAEs) | 30 days
  MAEs include stroke, cardiovascular death, new renal failure, endocarditis requiring surgery, and non-elective cardiovascular interventions due to device-related adverse events

SECONDARY OUTCOMES:
Acute procedural success | Immediately after procedure
  Successful in DragonFly-T implantation, and residual TR of 2+ or less at discharge. An echocardiography echocardiogram at 30 days can be accepted if the discharge image was not available or hard to interpret. A death before discharge or a re-operation of tricuspid valve prior to 30 days is defined as acute procedure failure
Acute device success | Immediately after procedure
  One or more DragonFly-T devices are successfully delivered and released, edge-to-edge leaflet repair confirmed by echocardiogram, and successfully withdrawal of the delivery catheter
Incidence of all-cause mortality and/or heart failure rehospitalization | 12 months
  Incidence of all-cause mortality and/or heart failure rehospitalization
Tricuspid regurgitation severity | 30 days, 6 months, 12 months
  Percentage of patients with tricuspid regurgitation of 2+ or less
Tricuspid regurgitation severity change | 30 days, 6 months, 12 months
  Percentage of patients with tricuspid regurgitation reduced by at least one grade
Change in 6 Minutes Walk Test | 30 days, 6 months, 12 months
  Improvement in 6 Minute Walk Test
Change in NYHA class | 30 days, 6 months, 12 months
  Improvement in New York Heart Association (NYHA) Function Class
Quality of life improvement | 30 days, 6 months, 12 months
  Improvement in quality of life (QoL) , as measured by the Kansas City Cardiomyopathy Questionnaire
Change in edema grading | 30 days, 6 months, 12 months
  Improvement in grading of edema，1-4 grade scale，higher scores mean worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jian'an Wang, MD,Phd, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No